CLINICAL TRIAL: NCT05267145
Title: The Protection of Blood Preservation Solution III on Erythrocytes in Intraoperative Blood Salvage During Cardiopulmonary Bypass
Brief Title: The Protection of ACD III on Erythrocytes in Intraoperative Blood Salvage During Cardiopulmonary Bypass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-0347
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-12

CONDITIONS: Red Blood Cell Disorder
Keywords: blood preservation solution III; intraoperative blood salvage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the blood storage bag contains blood preservation solution III (Experimental): a blood storage bag containing blood preservation solution III preserves the washed RBC
  Interventions: Combination Product: blood preservation solution III
- empty blood bag to store washed RBC (No Intervention): an empty blood storage bag preserves the washed RBC

INTERVENTIONS:
Combination Product: blood preservation solution III — Blood bag added blood preservation solution III
  Arms: the blood storage bag contains blood preservation solution III

SUMMARY:
To evaluate the effects of blood preservation solution III (sodium citrate, sodium dihydrogen phosphate, sodium citrate, glucose and adenine) in autologous blood recovery and storage bags on the metabolic morphological functions and characteristics of red blood cells in patients undergoing cardiac surgery supported by cardiopulmonary bypass

DETAILED DESCRIPTION:
Blood preservation solution III is a blood protective solution clinically used to store whole blood and red blood cells. It is a sterilized aqueous solution composed of sodium citrate dihydrogen phosphate sodium citrate glucose and adenine, in which glucose adenine can provide the required energy for stored RBC. Citric acid/sodium citrate buffer pair can adjust the pH of RBC suspension; Sodium dihydrogen phosphate can prevent RBC aggregation, provide phosphate for RBC energy metabolism, and slow down the decline rate of 2,3-DPG. Blood preservation solution III can reduce RBC destruction and protect its function. Therefore, this study aims to explore the effect of adding blood preservation solution III in blood storage bags on CPB Influence of autologous blood recovery RBC during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

Elective median incision for cardiac surgery under CPB ASAⅠ~Ⅲ Intraoperative blood recovery is pollution-free No blood system diseases, no red blood cell related diseases Preoperative blood routine examination showed no obvious abnormalities in blood coagulation function and biochemistry

Exclusion Criteria:

* Patients have malignant tumor Patients are complicated with systemic infectious disease Intraoperative blood loss is expected to be less than 200ml Patients receiving allogeneic red blood cells during operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
hemoglobin and free hemoglobin concentrations | up to 48 hours
  hemoglobin and free hemoglobin concentrations in both groups

SECONDARY OUTCOMES:
RBC morphology | autologous blood transfusion immediately, 24 hours, 48 hours
  erythrocyte morphology was observed by Rayner's staining and examined under microscope
Adenosine acid (ATP ADP AMP) content in RBC | autologous blood transfusion immediately, 24 hours, 48 hours
  the clarified supernatants were used for ATP, ADP, and AMP measurements with kits
2, 3-diphosphate (2,3-DPG) concentration | autologous blood transfusion immediately, 24 hours, 48 hours
  the cellular 2,3-DPG was analyzed fluorometrically with a kit

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China